CLINICAL TRIAL: NCT01638767
Title: Effect of Using the Nuvaring on the Level of Satisfaction, Stress on Users and on Coordinating In Vitro Fertilization (IVF) Cycles: Randomized Public Study
Brief Title: NuvaRing Versus Marvelon in the Coordination of In Vitro Fertilization Cycles
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty to recruit patient due to lack of eligible patient
Sponsor: Clinique Ovo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: OVO-10-03
Record Dates: First submitted 2012-07-06; First posted 2012-07-12 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Infertility
Keywords: In Vitro Fertilization long protocol; NuvaRing; Marvelon; In vitro fertilization
MeSH Terms: conditions — Infertility | interventions — Contraceptives, Oral; Desogestrel; Contraceptive Agents; Contraceptive Devices, Female; NuvaRing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NuvaRing (Experimental): Patients in the NuvaRing group will be inserting the vaginal ring for a period specified by the administrative nurse, ranging from 14 to 35 days.
  Interventions: Drug: Contraceptive, Vaginal ring
- Marvelon (Active Comparator): Patients on Marvelon will be taking the medication for a period ranging from 14 to 21 days. This period will be determined by the administrative nurse.
  Interventions: Drug: Contraceptives, Oral

INTERVENTIONS:
Drug: Contraceptives, Oral — 0.150 mg desogestrel and 0.030 mg ethinyl estradiol tablets, USP. One tablet per day at the same time each day, from the beginning of the menstrual cycle.
  Other Names: Marvelon
  Arms: Marvelon
Drug: Contraceptive, Vaginal ring — etogestrel/ ethinyl estradiol slow release vaginal ring (11.4 mg/2.6 mg) to deliver 120 mcg etonogestrel/15 mcg ethinyl estradiol per day
  Other Names: NuvaRing
  Arms: NuvaRing

SUMMARY:
Presently, a long protocol in an In Vitro Fertilization (IVF) cycle, patients need to take Marvelon, a drug that inhibits the follicular development at the beginning of the cycle in order to better control and also plan the onset of the ovary stimulation with gonadotropin.

Marvelon is taken daily as soon as menstruation starts for a period of 14 to 21 days. Ideally, it has to be taken at the same time everyday and not be forgotten. This may cause higher stress level for some users. Presently on the market, there is a ring-shaped contraceptive device inserted in the vagina at day 1 of the cycle called NuvaRing. The purpose of this device is similar to an oral contraceptive. However, the benefit of NuvaRing is that it can be left in place for a period of up to 35 days without any other manipulation and keep an adequate rate of hormone for contraception. Moreover, NuvaRing shows better hormone stability in the blood. Although the side effects and the benefits are comparable for the two treatments, some studies have shown that more patients would respect the treatment with NuvaRing and that the level of satisfaction would be higher in women using NuvaRing when contraception is needed.

The purpose of the study is to compare the rate of satisfaction as well as the level of stress in women using Marvelon daily or NuvaRing with single insertion in a long protocol. Moreover, this study allow us to verify if using NuvaRing, a vaginal contraceptive releasing constant daily doses for up to 35 days will allow us to facilitate the planning of In Vitro Fertilization cycles in long protocol.

DETAILED DESCRIPTION:
For the purpose of this randomized, controlled, open-label study, women will be selected from those undergoing in vitro fertilization treatments with a long protocol prescription. This study will compare two treatment groups, one using Marvelon, the other using the NuvaRing. Patients on Marvelon will be taking the medication for a period ranging from 14 to 21 days. This period will be determined by the administrative nurse. In contrast, patients in the NuvaRing group will be inserting the vaginal ring for a period specified by the administrative nurse, ranging from 14 to 35 days.

During the medical consultation, the couple will be assessed and a primary or secondary infertility diagnosis will be established. Before treatment starts, the couple will have to undergo a series of tests as per the standard of care in order to allow a diagnosis to be made and to determine whether In Vitro Fertilization is the right treatment. The couple will receive all the information they need on an In Vitro Fertilization cycle. If the patient is eligible for In Vitro Fertilization cycle according to initial assessment of the physician, the patient will be informed by the physician about the research project. After a period of consideration and once their questions have been answered, the couple will sign a consent form to start In Vitro Fertilization treatment under the study protocol

After signing the consent form, if the subject is eligible for the research project, the research nurse will meet with the patient. The study will be explained in detail and all questions will be answered. In addition, the nurse will record any information on the patient's medical history including medical history, medication and any previous surgery. The subject will be screened for eligibility prior to randomization. Once the subject is deemed eligible and is interested in participating in the study, the research nurse will meet with the subject in order to sign the informed consent form and to determine the randomization group she will be participating in. In order to determine which group will be allocated for a subject, a randomized envelope will be given to the patient containing the patient number will be opened to assign her to one of the two groups - either the Marvelon or the NuvaRing group. She will open it on site The randomization will be carried out using an envelope system to be identified initially by its randomization number. The envelopes will be prepared in advance in such a way that nobody can know their content.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form
* Age 18 or above at the time of selection
* In Vitro Fertilization referral
* Complete and normal pre-In Vitro Fertilization check-up
* Long protocol prescription
* No previous participation in the project during a previous cycle

Exclusion Criteria:

* Simultaneous participation in another interventional research project
* Contraindications of being pregnant or carrying a pregnancy to full term
* Contraindications of taking standard medication for long protocol
* Contraindications of taking Marvelon or using NuvaRing (Uncontrolled high blood pressure, uncontrolled diabetes, active hepatic infection, benign or malignant hepatic tumors, diagnosed breast cancer, diagnosed or suspected estrogen-dependant neoplasia, ocular or suspected lesion, history of thrombophlebitis, cardiac arrest, coronary heart disease.)
* Patient presenting vaginal abnormalities could be unable to insert the NuvaRing
* Cervicitis, vaginitis, erosio portionis bleeding, cervical prolapse, cystocele, rectocele, severe or chronic constipation, dyspareunia or other problems with sexual intercourse
* Patient having received research medication 30 days before visit 1
* Patient is unable to communicate adequately with researchers
* Patient is incapable of giving informed consent
* Any ovarian or abdominal abnormalities could interfere with an adequate sonographic evaluation
* Use of the following medication:
* Clonidine
* Anticoagulants (before the anovulant pre-treatment)
* Anticonvulsants
* Oral or insulin hypoglycemia drugs
* Hypertension drugs (beta blockers)
* Aminocaproic acid
* Beta mimetics (isoproterenol)
* Prednisone
* Ciclosporin
* Meperidine
* Phenothiazine and reserpine
* Chlordiazepoxide, Lorazepam, Oxazepam, Diazepam (during the anovulant pre-treatment)
* Theophylline
* Clomipramine
* Vitamin B12
* Hypericum perforatum-based products

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The level of satisfaction in patients in relation to contraceptive medication | From date of the beginning of the In Vitro Fertilization cycle until the end of the cycle, assesses up to 65 days.
The level of stress experienced by patients in relation to contraceptive medication | From date of the beginning of the In Vitro Fertilization cycle until the end of the cycle, assesses up to 65 days.
Patient's adherence to the treatment | From date of the beginning of the In Vitro Fertilization cycle until the end of the cycle, assesses up to 65 days.
The number of patients who had bleeding during their contraceptive treatment | From date of the beginning of the In Vitro Fertilization cycle until the end of the cycle, assesses up to 65 days.
The level of satisfaction among administrative nurses in regards to planning the cycle. | From date of the beginning of the In Vitro Fertilization cycle until the end of the cycle, assesses up to 65 days.

SECONDARY OUTCOMES:
The number of follicles at the last sonogram before the Human chorionic gonadotropin (hCG) injection | At time of the last sonogram before the Human chorionicgonadotropin (hCG) injection, approximately 20 days
The presence of cysts (diameter ≥ 15 mm) | From date of the beginning of the In Vitro Fertilization cycle until the end of the cycle, assesses up to 65 days.
The number of mature ova recovered | At the time of ova retrieval, approximately 20 days
The number of usable embryos | From the time of ova retrieval until the time of embryo transfer, up to 5 days.
The pregnancy rates | At the time of the pregnancy test, approximately 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kadoch, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

REFERENCES:
- [Background] Timmer CJ, Mulders TM. Pharmacokinetics of etonogestrel and ethinylestradiol released from a combined contraceptive vaginal ring. Clin Pharmacokinet. 2000 Sep;39(3):233-42. doi: 10.2165/00003088-200039030-00005. PMID 11020137
- [Background] Roumen FJ, Apter D, Mulders TM, Dieben TO. Efficacy, tolerability and acceptability of a novel contraceptive vaginal ring releasing etonogestrel and ethinyl oestradiol. Hum Reprod. 2001 Mar;16(3):469-75. doi: 10.1093/humrep/16.3.469. PMID 11228213
- [Background] Novak A, de la Loge C, Abetz L, van der Meulen EA. The combined contraceptive vaginal ring, NuvaRing: an international study of user acceptability. Contraception. 2003 Mar;67(3):187-94. doi: 10.1016/s0010-7824(02)00514-0. PMID 12618252